CLINICAL TRIAL: NCT01234311
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study of Tasquinimod in Men With Metastatic Castrate Resistant Prostate Cancer
Brief Title: A Study of Tasquinimod in Men With Metastatic Castrate Resistant Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Active Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10TASQ10
Record Dates: First submitted 2010-11-01; First posted 2010-11-04 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tasquinimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo
- tasquinimod (Experimental): Tasquinimod up to a maximum maintenance dose of 1 mg once daily, administrated orally (capsule)
  Interventions: Drug: tasquinimod

INTERVENTIONS:
Drug: tasquinimod — Tasquinimod up to a maximum maintenance dose of 1 mg once daily, administrated orally (capsule)
  Other Names: ABR-215050
  Arms: tasquinimod
Drug: Placebo
  Arms: placebo

SUMMARY:
This is a Phase 3 randomized, double blind, placebo controlled study of tasquinimod in asymptomatic to mildly symptomatic patients with metastatic CRPC to confirm the effect of tasquinimod on delaying disease progression compared with placebo.

Approximately 1200 eligible patients with metastatic CRPC will be randomly assigned in a 2:1 ratio to 1 of 2 treatment groups: Treatment Group A (tasquinimod 0.25, 0.5, or 1 mg/day; n=800) or Treatment Group B (placebo; n=400).

DETAILED DESCRIPTION:
This is a Phase 3 randomized, double blind, placebo controlled study of tasquinimod in asymptomatic to mildly symptomatic patients with metastatic CRPC to confirm the effect of tasquinimod on delaying disease progression compared with placebo.

Approximately 1200 eligible patients with metastatic CRPC will be randomly assigned in a 2:1 ratio to 1 of 2 treatment groups: Treatment Group A (tasquinimod 0.25, 0.5, or 1 mg/day; n=800) or Treatment Group B (placebo; n=400).

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years at the time of signing the informed consent form. For patients in Taiwan the minimum age is 20 years.
2. Histologically confirmed diagnosis of adenocarcinoma of the prostate.
3. Evidence of bone metastatic disease on radiographic examination, whether from bone scan or other imaging modality.
4. Castrate levels of serum testosterone (≤50 ng/dL or 1.7 nmol/L).
5. Evidence of progressive disease.
6. Karnofsky score ≥70%.
7. Meet screening laboratory values as specified in thr protocol.
8. If sexually active with partner of childbearing potential, patient will agree to use adequate contraceptive methods (barrier contraceptive with spermicide or vasectomy) while on study drug. The adequate contraceptive method should be continued for 14 days after the patient stops taking study drug.
9. No evidence (within 5 years) of prior malignancies (except successfully treated basal cell or squamous cell carcinoma of the skin).
10. Able to swallow and retain oral medication.
11. Able to adhere to the study visit schedule and other protocol requirements.
12. Ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to cooperate with the investigator and to comply with the requirements of the entire study.
13. Able (or patient's legal guardian, if applicable) to sign and date the written informed consent after being informed of the full nature and purpose of the study, including possible risks and side effects, and given ample time and opportunity to read and understand this information.

Exclusion Criteria:

1. Prior cytotoxic chemotherapy for the treatment of prostate ca within 2 years or within 4 weeks for Estracyt (estramustine) prior to study treatment.
2. Previous anticancer therapy using radiation, biologics or vaccines, including abiraterone, TAK-700 (Orteronel), or MDV3100 within 4 weeks prior or sipuleucel-T (Provenge) within 2 weeks prior to the start of study treatment. If radiation therapy is applied after baseline scan, a new baseline scan needs to be done at least 4 weeks after the radiation therapy.
3. Previous therapy with antiandrogens within 4 weeks (within 6 weeks for bicalutamide eg, Casodex®) prior to study treatment.
4. Concurrent use of other anticancer agents or treatments, with the following exceptions:

   • Ongoing treatment with luteinizing hormone-releasing hormone agonists or antagonists, denosumab (Prolia) or bisphosphonate (eg, zoledronic acid) is allowed. Ongoing treatment should be kept at a stable schedule; however, if medically required, a change of dose, compound, or both is allowed.
5. Any treatment modalities involving major surgery within 4 weeks prior to the start of study treatment.
6. Prostate ca pain that requires ongoing treatment with narcotic analgesics or warrants the initiation of radio- or chemotherapy.
7. Ongoing treatment with warfarin unless the international normalized ratio (INR) is well controlled and below 4 (Section 4.6.8.1).
8. Maintenance treatment with corticosteroids corresponding to a prednisolone or prednisone dose above 10 mg/day. The dose must have been stable for at least 5 days.
9. Systemic exposure to ketoconazole or other strong cytochrome P450 (CYP) 3A4 isozyme inhibitors or inducers within 14 days prior to the start of study treatment. Systemic exposure to amiodarone is not allowed within 1 year prior to the start of study treatment.
10. Ongoing treatment with sensitive CYP1A2 substrate or CYP1A2 substrate with narrow therapeutic range at the start of study treatment.
11. Ongoing treatment with CYP3A4 substrate with narrow therapeutic range at the start of study treatment.
12. Simultaneous participation in any other study involving treatment with investigational drugs or having received treatment with investigational drugs less than 4 weeks prior to the start of study treatment.
13. Myocardial infarction, percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass graft, class III/IV congestive heart failure, cerebrovascular accident, transient ischemic attack, or limb claudication at rest, within 6 months prior to start of study treatment and ongoing symptomatic dysrhythmias, unstable angina, uncontrolled hypertension, and uncontrolled atrial or ventricular arrhythmias.
14. History of pancreatitis.
15. Known brain or epidural metastases.
16. Known positive serology for HIV (patients with known history of HIV will be excluded because of potential for unforeseen toxicity and morbidity in an immunocompromised host).
17. Chronic hepatitis with advanced, decompensated hepatic disease or cirrhosis of the liver or history of a chronic viral hepatitis or known viral hepatitis carrier (patients who have recovered from hepatitis will be allowed to enter the study).
18. Patients with active tuberculosis (TB), or with known, untreated latent TB. (Country-specific TB therapy should have been given for at least 30 days prior to the start of study treatment and the patient should intend to complete the entire course of that therapy.)
19. Any condition, including other active or latent infections, medical or psychiatric conditions, or the presence of laboratory abnormalities, which could confound the ability to interpret data from the study or places the patient at unacceptable risk if he participates in the study.
20. Any patient who in the opinion of the investigator should not participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1245 (Actual)
Dates: Start 2011-03; Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study of Tasquinimod in Men with Metastatic Castrate Resistant Prostate Cancer | 5 years
  The primary endpoint is progression-free survival (PFS) defined as the time from the date of randomization to the date of radiological progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Carducci, MD, Principal Investigator — Johns Hopkins Kimmel Cancer Center, Baltimore, MD
Locations (204):
- United States (34):
  - Tucson, Arizona
  - Oxnard, California
  - Santa Monica, California
  - Santa Rosa, California
  - Wellington, Florida
  - Atlanta, Georgia
  - Meridian, Idaho
  - Melrose Park, Illinois
  - Park Ridge, Illinois
  - Jeffersonville, Indiana
  - Baltimore, Maryland
  - Rockville, Maryland
  - Boston, Massachusetts
  - Jefferson City, Missouri
  - Las Vegas, Nevada
  - Hackensack, New Jersey
  - Lawrenceville, New Jersey
  - Buffalo, New York
  - Poughkeepsie, New York
  - Concord, North Carolina
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Springfield, Oregon
  - Bala-Cynwyd, Pennsylvania
  - Lancaster, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Myrtle Beach, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Salt Lake City, Utah
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Salem, Virginia
  - Burien, Washington
- Argentina (3):
  - Buenos Aires
  - Santa Rosa
  - Venado Tuerto
- Australia (6):
  - Camperdown, New South Wales
  - Coffs Harbour, New South Wales
  - Darlinghurst, New South Wales
  - Tweed Heads, New South Wales
  - Richmond, Victoria
  - Subiaco, Western Australia
- Belgium (4):
  - Brussels
  - Ghent
  - Kortrijk
  - Liège
- Brazil (13):
  - Botucatu, Sao Paulo
  - Cachoeiro de Itapemirim - ES
  - Curitiba, Parana
  - Florianópolis
  - Juiz de Fora, Minas Gerais
  - Mogi Das Cruzes, Sao Paulo
  - Natal, Rio Grande Do Norte
  - Passo Fundo
  - Porto Alegre, RS
  - Rio de Janeiro
  - Salvador/BA
  - São Paulo
  - Volta Redonda - RJ
- Bulgaria (4):
  - Pleven
  - Plovdiv
  - Sofia
  - Varna
- Canada (5):
  - Kelowna, British Columbia
  - Victoria, British Columbia
  - Brantford, Ontario
  - North York, Ontario
  - Oakville, Ontario
- Chile (3):
  - Santiago
  - Temuco
  - Viña del Mar
- China (5):
  - Beijing
  - Chengdu
  - Shanghai
  - Shantou
  - Wuhan
- Colombia (2):
  - Bogotá
  - Cali
- Czechia (4):
  - Nový Jičín
  - Olomouc
  - Prague
  - Ústí nad Labem
- Tartu, Estonia
- France (8):
  - Angers
  - Cannes
  - Marseille
  - Montpellier
  - Paris
  - Pierre-Bénite
  - Rennes
  - Suresnes
- Germany (10):
  - Cologne
  - Dresden
  - Hamburg
  - Mannheim
  - Marburg
  - München
  - Münster
  - Nürtingen
  - Tübingen
  - Weiden
- Greece (3):
  - Athens
  - Pátrai
  - Thessaloniki
- Pune, India
- Israel (7):
  - Beersheba
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
  - Ẕerifin
- Italy (8):
  - Cremona
  - Lecco
  - Meldola
  - Milan
  - Padua
  - Ravenna
  - Roma
  - Torino
- Latvia (2):
  - Liepāja
  - Riga
- Lebanon (2):
  - Beirut
  - Bsalîm
- Lithuania (2):
  - Kaunas
  - Vilnius
- Mexico (5):
  - Chihuahua, Chih.
  - Culiacan, Sinaloa
  - Leon, GTO
  - Puebla City
  - Zapopan, Jalisco
- Netherlands (5):
  - Amsterdam
  - Groningen
  - Leiden
  - Nijmegen
  - Tilburg
- New Zealand (4):
  - Christchurch
  - Nelson
  - Palmerston North
  - Tauranga
- Panama City, Panama
- Arequipa, Peru
- Poland (6):
  - Bialystok
  - Lodz
  - Mysłowice
  - Poznan
  - Warsaw
  - Wroclaw
- Romania (7):
  - Baia Mare
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Ploieşti
  - Suceava
  - Timișoara
- Russia (6):
  - Moscow
  - Novosibirsk
  - Omsk
  - Saint Petersburg
  - Vladimir
  - Yekaterinburg
- Slovakia (2):
  - Bratislava
  - Trenčín
- South Korea (2):
  - Gwangju
  - Seoul
- Spain (10):
  - Seville, Andalusia
  - Zaragoza, Aragon
  - Santander, Cantabria
  - Sabadell, Catalonia
  - Alcorcón, Madrid, Communidad de
  - Pamplona, Navarre
  - Oviedo, Principality of Asturias
  - Barcelona
  - San Sebastián de los Reyes
  - Valencia
- Sweden (3):
  - Gothenburg
  - Karlstad
  - Stockholm
- Taiwan (4):
  - Kaohsiung City
  - Taichung
  - Taipei
  - Taoyuan District
- Istanbul, Turkey (Türkiye)
- Ukraine (11):
  - Chernivtsi
  - Dnipropetrovsk
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kyiv
  - Lutsk
  - Lviv
  - Odesa
  - Uzhhorod
  - Zaporizhzhya
- United Kingdom (9):
  - Birmingham
  - Chichester
  - Leeds
  - London
  - Northwood
  - Nottingham
  - Oxford
  - Scunthorpe
  - Sutton

REFERENCES:
- [Derived] Armstrong AJ, Anand A, Edenbrandt L, Bondesson E, Bjartell A, Widmark A, Sternberg CN, Pili R, Tuvesson H, Nordle O, Carducci MA, Morris MJ. Phase 3 Assessment of the Automated Bone Scan Index as a Prognostic Imaging Biomarker of Overall Survival in Men With Metastatic Castration-Resistant Prostate Cancer: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2018 Jul 1;4(7):944-951. doi: 10.1001/jamaoncol.2018.1093. PMID 29799999
- [Derived] Sternberg C, Armstrong A, Pili R, Ng S, Huddart R, Agarwal N, Khvorostenko D, Lyulko O, Brize A, Vogelzang N, Delva R, Harza M, Thanos A, James N, Werbrouck P, Bogemann M, Hutson T, Milecki P, Chowdhury S, Gallardo E, Schwartsmann G, Pouget JC, Baton F, Nederman T, Tuvesson H, Carducci M. Randomized, Double-Blind, Placebo-Controlled Phase III Study of Tasquinimod in Men With Metastatic Castration-Resistant Prostate Cancer. J Clin Oncol. 2016 Aug 1;34(22):2636-43. doi: 10.1200/JCO.2016.66.9697. Epub 2016 Jun 13. PMID 27298414